CLINICAL TRIAL: NCT06563531
Title: Are Elastic Restraints Still Necessary in Improved Rehabilitation Programs After Hip and Knee Prosthetic Surgery?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Pasteur Lanroze (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022-04-CPL
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Arthroplasty Complications
Keywords: hip replacement surgery; knee replacement surgery; thromboprophylaxis; elastic compression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Elastic compression (Active Comparator)
  Interventions: Procedure: Pharmacological thromboprophylaxis and elastic compression
- No elastic compression (Experimental)
  Interventions: Procedure: Pharmacological thromboprophylaxis without elastic compression

INTERVENTIONS:
Procedure: Pharmacological thromboprophylaxis and elastic compression — Patients benefit from thromboembolism prevention through pharmacological thromboprophylaxis and elastic restraint after total hip or knee arthroplasty.
  Arms: Elastic compression
Procedure: Pharmacological thromboprophylaxis without elastic compression — Patients benefit from thromboembolism prevention through pharmacological thromboprophylaxis only after total hip or knee arthroplasty.
  Arms: No elastic compression

SUMMARY:
Venous thrombosis and pulmonary embolism are considered serious and potentially preventable complications of hip and knee replacement surgery. The risks of thrombosis must be weighed against the risks associated with preventive measures, both mechanical and pharmacological. Modern medicine is now questioning the use of elastic restraints in surgery. Several studies have investigated the benefits of using restraints to prevent thromboembolic events. These studies have shown no additional benefit from the use of compression stockings in thromboembolism prevention. To the best of our knowledge, no orthopedic study has investigated the non-inferiority of pharmacological treatment compared with elastic compression devices, specifically in knee and hip surgery. The aim of this multicenter, prospective, randomized study is to investigate whether pharmacological prophylaxis alone is non-inferior to pharmacological and mechanical prophylaxis (using restraints) of peripheral venous thrombosis or pulmonary embolism up to 90 days after prosthetic surgery.

ELIGIBILITY:
Inclusion Criteria:

* first line and non-traumatic total hip or knee arthroplasty
* Patient included in an Enhanced Rehabilitation after Surgery (ERS) or "fast-track" protocol, or scheduled as an outpatient.

Exclusion Criteria:

* Patient requiring long-term anticoagulation for pre-existing co-morbidity
* Patients with coagulation disorders (hypercoagulability)
* Patient undergoing thrombogenic pharmacological treatment
* History of obliterative arteriopathy of the lower limbs
* Arterial disease
* Obesity
* Heart failure
* Chronic bronchopneumopathy
* Lymphedema
* Chronic inflammatory disease
* Permanent wearing of elastic restraints
* Proximal or distal arterial bypass surgery
* Creatinine clearance < 15 ml/min
* Inability to give consent
* Revision surgery for hip or knee prosthesis
* Metastatic cancer
* Life expectancy less than 3 months
* Allergy to socks or compression stockings
* Patients presenting one or more exclusion criteria for the fast-track protocol (severe or poorly-balanced associated conditions such as diabetes or immunodepression, inability to contact the doctor or hospital department if necessary, pre-operative ASA score greater than or equal to 4).
* Adults under guardianship or curatorship
* Vulnerable persons in accordance with article L1121-6 of the CSP (French Public Health Code)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1274 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
incidence of venous thromboembolic events | day 1 ; day 21 ; day 90
  Evaluation of venous thromboembolic events (symptomatic deep vein thrombosis, fatal or non-fatal pulmonary embolism).

SECONDARY OUTCOMES:
Quality of life evaluation | day 1 ; day 21 ; day 90
  Quality of life will be evaluated by EQ-5D-5L questionnaire : 5 questions with a Likert scale from 0 (no symptoms) to 4 (extreme symptoms), with a final result from 0 to 20.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Pasteur Lanroze, Brest, France

IPD SHARING:
Plan to Share IPD: No